CLINICAL TRIAL: NCT05745246
Title: Firefighters Preventing Cancer: Cluster Randomized Trial of an Online Training Program for Cancer Prevention Behaviors in Volunteer Firefighters
Brief Title: Firefighters Preventing Cancer Online Training Program
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IWK Health Centre (Other)
Collaborators: Canadian Association of Fire Chiefs (Unknown); Laval University (Other)
Responsible Party: Principal Investigator, Patrick J. McGrath, Principle Investigator, IWK Health Centre
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 1028192
Record Dates: First submitted 2023-02-16; First posted 2023-02-27 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Cancer Prevention
Keywords: Firefighter; Cancer; Decontamination; Exposure
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: This study is a two-arm, feasibility, Cluster Randomized Trial (CRT).
Who Masked: Investigator, Outcomes Assessor
Masking Description: Since this study is a Cluster Randomized Trial (CRT), first, Departments will be recruited and randomized to the treatment arm or the control arm, with a 1:1 allocation ratio stratified by region. The randomization sequence will be generated by a trained person that is not related to the study participants in any way. The investigators and study staff will be blinded to the randomization sequence until the end of the study. Participant randomization will be performed in REDCap. REDCap maintains an automated audit trail which includes the assigned study identification number, treatment allocation, and date and time of the allocation assignment.
  Once a department is recruited and assigned to a study group, all the members in that department will be assigned to the same group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): This arm will receive the online e-health intervention for six months.
  The intervention consists of three sections:
  1. a novel health information strategy, 90SecondFire Cancer health letters
  2. a brief on-line course
  3. a problem-solving asynchronous bulletin board to mobilize existing knowledge
  Interventions: Behavioral: e-health training program
- waitlist control group (No Intervention): This group will be placed on a waitlist and will receive the online treatment program after six months.

INTERVENTIONS:
Behavioral: e-health training program — 1. Health letters, 44 issues of 90SecondFire Cancer health letters delivered twice a week during six months to firefighters by text or email
  2. A problem-solving asynchronous chat room which encourages mutual support and exchange of ideas via a closed asynchronous bulletin board for peer-to-peer support
  3. A brief 45-minute pre-recorded online course; it is intended as a summative exercise rather than providing new information.
  Arms: Intervention Group

SUMMARY:
The goal of this two-arm, Cluster Randomized Trial is to evaluate an e-health training program for volunteer firefighters to reduce their risk of exposures to carcinogens and to increase their understanding and intentions of behavior towards cancer prevention. One arm will receive an online e-health intervention for six months and the other arm will be considered as a waitlist control group which will be placed on a waitlist and receive the online treatment program some months later.

The project aims to evaluate the firefighters by measurement of current behavior, perceived importance, future behavioral intentions and perceived barriers for implementing decontamination behaviors at baseline, after the intervention and after 3-month follow-up before and after the intervention.

The intervention consists of three components:

1. a novel health information strategy, 90SecondFire Cancer health letters
2. a brief on-line course
3. a problem-solving asynchronous bulletin board to mobilize existing knowledge

DETAILED DESCRIPTION:
Firefighters face a serious risk of exposure to carcinogens from products of combustion. Modern materials burn hotter and may be even more toxic than older wood construction. Preventing the increased risk of cancer in volunteer firefighters has raised attention as they are more vulnerable to carcinogen exposure.

The goal of this two-arm, Cluster Randomized Trial is to evaluate an e-health training program for volunteer firefighters to reduce their risk of exposures to carcinogens and to increase their understanding and intentions of behavior towards cancer prevention. One arm will receive an online e-health intervention for six months and the other arm will be considered as a waitlist control group which will be placed on a waitlist and receive the online treatment program some months later. Up to 800 volunteer firefighters from approximately 40 volunteer fire departments in Canada will be recruited for both arms.

The project aims to evaluate the firefighters by measurement of current behavior, perceived importance, future behavioral intentions and perceived barriers for implementing decontamination behaviors at baseline, after the intervention and after 3-month follow-up through an online validated survey: Firefighter Exposure to Carcinogens Scale (FECS).

The intervention consists of three components:

1. a novel health information strategy, 90SecondFire Cancer health letters
2. a brief on-line course
3. a problem-solving asynchronous bulletin board to mobilize existing knowledge

ELIGIBILITY:
Inclusion Criteria:

Departments will be screened to meet the following criteria

1. Be a Volunteer Department
2. Be located in Canada
3. Consent to participate in the study via the Chief or delegate

Participant in the CRT study must meet all the following criteria to be eligible to proceed with the study:

1. Be a volunteer firefighter
2. Working for an all-volunteer fire department that has joined the study
3. Live in Canada
4. Has access to internet
5. Be able to read, write and understand English or French
6. Consent to participate in the study

Exclusion Criteria:

The exclusion for Departments

1. Not a volunteer Department in other words to be a composite department with some volunteers and some career fire fighters or a department that has not joined the study
2. Not located in Canada
3. Not Consent to be in the study via the Chief or delegate

Any of the following criteria will exclude individuals from proceeding to consent:

1. NOT a volunteer firefighter
2. Working for a composite department with some volunteers and some career fire fighters or a department that has not joined the study
3. Does NOT live in Canada
4. Does not have access to internet
5. Is NOT able to read, write and understand English or French
6. Does NOT consent to participate in the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 179 (Actual)
Dates: Start 2023-02-13 (Actual); Primary Completion 2024-10-30 (Actual); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Volunteer Firefighters' Intention to engage in reducing exposure and undertaking decontamination behaviour | Baseline, After 6 month intervention and 3-month follow-up
  In order to measure the changes in firefighter's intention during the study, the data will be collected by an online survey: Firefighter Exposure to Carcinogens Scale. The dimensions will be rated on a Likert scale. min :0 Max 4 ; The higher score does not mean a better outcome.

SECONDARY OUTCOMES:
Volunteer Firefighters' practice and perceived importance towards reducing exposure and undertaking decontamination behavior for cancer prevention | Baseline, After 6 month intervention and 3-month follow-up
  The data will be collected by an online survey: Firefighter Exposure to Carcinogens Scale . The dimensions will be rated on a Likert scale. min :0 Max 4 ; The higher score does not mean a better outcome.
Volunteer firefighters' and their departments' perceived barriers in the development of reducing exposure and undertaking decontamination behaviors | Baseline, After 6 month intervention and 3-month follow-up
  The data will be collected by an online survey: Firefighter Exposure to Carcinogens Scale . The dimensions will be rated on a a Likert scale. min :0 Max 4 ; The higher score does not mean a better outcome.
Comparing and detecting any association between the regular volunteer firefighters and the management team towards cancer prevention | Baseline, After 6 month intervention and 3-month follow-up
  The data will be collected by an online survey: Firefighter Exposure to Carcinogens Scale . The dimensions will be rated on a Likert scale. min :0 Max 4 ; The higher score does not mean a better outcome.
Comparing characteristics of different volunteer Departments (Clusters) such as size and location of Department in terms of their future intention, current practice and perceived importance towards cancer prevention | Baseline, After 6 month intervention and 3-month follow-up
  The data will be collected by an online survey: Firefighter Exposure to Carcinogens Scale . The dimensions will be rated on a Likert scale. min :0 Max 4 ; The higher score does not mean a better outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- IWK Health Centre, Halifax, Nova Scotia, Canada